CLINICAL TRIAL: NCT05181085
Title: A Phase 1, First Time in Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NST 6179 in Healthy Subjects
Brief Title: Study of NST-6179 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NorthSea Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NST-6179-01
Record Dates: First submitted 2021-08-30; First posted 2022-01-06 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Short Bowel Syndrome; Parenteral Nutrition Associated Liver Disease
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NST 6179 (Active Comparator): double blind, single ascending and multiple ascending dose, sequential group design
  Interventions: Drug: NST 6179
- Placebo (Placebo Comparator): matched placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NST 6179 — orally administered, fully synthetic medium chain fatty acid (MCFA) analogue
  Arms: NST 6179
Drug: Placebo — inactive analogue
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo controlled, single and multiple oral dose study to assess safety and tolerability of single and multiple doses of NST-6179 in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 65 years of age, inclusive.
2. Body mass index between 18.0 and 32.0 kg/m^2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and/or check in as assessed by the investigator (or designee).
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
5. Able to comprehend and willing to sign an ICF and to abide by the study restrictions

Exclusion Criteria (additional criteria available):

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
3. Any of the following:

   1. QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 ms confirmed by repeat measurement.
   2. QRS duration > 110 ms confirmed by repeat measurement.
   3. PR interval > 220 ms confirmed by repeat measurement.
   4. findings which would make QTc measurements difficult or QTc data uninterpretable.
   5. history of additional risk factors for torsades de pointes (eg, heart failure, hypokalaemia, family history of long QT syndrome).
4. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the investigator (or designee).
5. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the investigator (or designee).
6. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing.
7. Vegetarians, vegans, and/or unable to consume the high fat breakfast (subjects participating in a food effect evaluation only).
8. History of alcoholism or drug/chemical abuse within 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Ltd, Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Dose Placebo: Participants in Part A randomised to receive a single dose of placebo.
- Single Dose 50 mg NST-6179: Participants in Part A randomised to receive a single dose of 50 mg NST-6179.
- Single Dose 200 mg NST-6179: Participants in Part A randomised to receive a single dose of 200 mg NST-6179.
- Single Dose 400 mg NST-6179: Participants in Part A randomised to receive a single dose of 400 mg NST-6179.
- Single Dose 600 mg NST-6179: Participants in Part A randomised to receive a single dose of 600 mg NST-6179.
- Single Dose 1000 mg NST-6179: Participants in Part A randomised to receive a single dose of 1000 mg NST-6179.
- Multiple Dose Placebo: Participants in Part B randomised to receive multiple doses of placebo.
- Multiple Dose 200 mg NST-6179 (QD): Participants in Part B randomised to receive multiple doses of 200 mg NST-6179 (QD).
- Multiple Dose 400 mg NST-6179 (QD): Participants in Part B randomised to receive multiple doses of 400 mg NST-6179 (QD).
- Multiple Dose 1000 mg NST-6179 (QD): Participants in Part B randomised to receive multiple doses of 1000 mg NST-6179 (QD).
Period: Overall Study
Arm/Group | Single Dose Placebo | Single Dose 50 mg NST-6179 | Single Dose 200 mg NST-6179 | Single Dose 400 mg NST-6179 | Single Dose 600 mg NST-6179 | Single Dose 1000 mg NST-6179 | Multiple Dose Placebo | Multiple Dose 200 mg NST-6179 (QD) | Multiple Dose 400 mg NST-6179 (QD) | Multiple Dose 1000 mg NST-6179 (QD)
Started | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose Placebo | Single Dose 50 mg NST-6179 | Single Dose 200 mg NST-6179 | Single Dose 400 mg NST-6179 | Single Dose 600 mg NST-6179 | Single Dose 1000 mg NST-6179 | Multiple Dose Placebo | Multiple Dose 200 mg NST-6179 (QD) | Multiple Dose 400 mg NST-6179 (QD) | Multiple Dose 1000 mg NST-6179 (QD) | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 70
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 3 | 2 | 2 | 3 | 3 | 4 | 0 | 29
  Male | 6 | 3 | 1 | 3 | 4 | 4 | 3 | 5 | 4 | 8 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 9 | 6 | 5 | 6 | 5 | 6 | 6 | 7 | 8 | 7 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AEs and SAEs Following Administration of NST 6179
Description: Assessment of number of participants with AEs and SAEs to determine safety profile
Time Frame: From screening to 14 days post final dose, up to 4 weeks.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Placebo | Single Dose 50 mg NST-6179 | Single Dose 200 mg NST-6179 | Single Dose 400 mg NST-6179 | Single Dose 600 mg NST-6179 | Single Dose 1000 mg NST-6179 | Multiple Dose Placebo | Multiple Dose 200 mg NST-6179 (QD) | Multiple Dose 400 mg NST-6179 (QD) | Multiple Dose 1000 mg NST-6179 (QD)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8
Participants
  Overall TEAEs | 4 | 2 | 2 | 2 | 2 | 2 | 2 | 5 | 6 | 5
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mild TEAEs | 4 | 2 | 2 | 2 | 2 | 1 | 2 | 5 | 5 | 5
  Moderate TEAEs | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 1
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Overall treatment-related TEAEs | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5 | 5
  Mild treatment-related TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 4
  Moderate treatment-related TEAEs | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1

2. Secondary Outcome: Peak Plasma Concentration (Cmax) of NST 6179
Description: Measure of peak plasma concentration of NST 6179 after dose on Day 1
Time Frame: Day 1
Population: PK population (all subjects who received NST-6179)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Single Dose 50 mg NST-6179 | Single Dose 200 mg NST-6179 | Single Dose 400 mg NST-6179 | Single Dose 600 mg NST-6179 | Single Dose 1000 mg NST-6179 | Multiple Dose 200 mg NST-6179 (QD) | Multiple Dose 400 mg NST-6179 (QD) | Multiple Dose 1000 mg NST-6179 (QD)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8
ng/mL | 1100 (54.7) | 4880 (49.9) | 13200 (29.2) | 18300 (33.7) | 27200 (33.7) | 5690 (51.0) | 10500 (60.4) | 29100 (25.3)

3. Secondary Outcome: Peak Plasma Concentration (Cmax) of NST 6179
Description: Measure of peak plasma concentration of NST 6179 after dose on Day 14
Time Frame: Day 14
Population: PK population (all subjects who received NST-6179)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Multiple Dose 200 mg NST-6179 (QD) | Multiple Dose 400 mg NST-6179 (QD) | Multiple Dose 1000 mg NST-6179 (QD)
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 6920 (28.0) | 10000 (34.9) | 31800 (39.9)

4. Other Pre Specified Outcome: NST 6179 Concentrations and QT Interval
Description: assess for correlation of potential cardiotoxicity by looking at PK of NST 6179 and ECG results collected
Time Frame: From screening to 14 days post final dose, up to 4 weeks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From screening to 14 days post final dose, up to 4 weeks.
Description: Reporting through regular investigator assessment.
Arm/Group | Single Dose Placebo | Single Dose 50 mg NST-6179 | Single Dose 200 mg NST-6179 | Single Dose 400 mg NST-6179 | Single Dose 600 mg NST-6179 | Single Dose 1000 mg NST-6179 | Multiple Dose Placebo | Multiple Dose 200 mg NST-6179 (QD) | Multiple Dose 400 mg NST-6179 (QD) | Multiple Dose 1000 mg NST-6179 (QD)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/10 | 2/6 | 2/6 | 2/6 | 2/6 | 2/6 | 2/6 | 5/8 | 6/8 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose Placebo (N=10) | Single Dose 50 mg NST-6179 (N=6) | Single Dose 200 mg NST-6179 (N=6) | Single Dose 400 mg NST-6179 (N=6) | Single Dose 600 mg NST-6179 (N=6) | Single Dose 1000 mg NST-6179 (N=6) | Multiple Dose Placebo (N=6) | Multiple Dose 200 mg NST-6179 (QD) (N=8) | Multiple Dose 400 mg NST-6179 (QD) (N=8) | Multiple Dose 1000 mg NST-6179 (QD) (N=8)
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site irritation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Micturition frequency decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT05181085/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT05181085/SAP_001.pdf